CLINICAL TRIAL: NCT05909865
Title: PRedIcting MEniscal Tears Outcomes After Physical Therapy Treatment (the PRIME Study): a Multivariable Prediction Model Development Study
Brief Title: PRedIcting MEniscal Tears Outcomes After Physical Therapy Treatment
Acronym: PRIME
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial support for the project has been discontinued.
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Collaborators: Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario La Princesa (Unknown); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Principe de Asturias (Other); Hospital Universitario de Fuenlabrada (Other); Hospital Universitario Infanta Leonor - Vallecas/H. Virgen de la Torre (Unknown)
Responsible Party: Principal Investigator, Rubén Fernández Matías, Principal Investigator, Hospital Universitario Fundación Alcorcón
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/67
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Meniscus Tear
Keywords: Physical therapy; Therapeutic resistance exercise; Education; Prediction model
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study will be a non-controlled multicenter clinical trial with the main aim of developing a multivariable prediction model of the improvements after a physical therapy treatment based on exercise and education.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic exercise plus education (Experimental): The treatment will consist of a progressive resistance exercise program along with education.
  Interventions: Other: Therapeutic resistance exercise; Other: Education

INTERVENTIONS:
Other: Therapeutic resistance exercise — Therapeutic exercise program based on individualized progressive resistance exercises performed during 3 months at home, with a frequency of 1-3 sessions per week at the hospital.
Other: Education — Education applied during all the therapeutic process, focusing on diverting the patient's attention away from the structural lesion, explaining the relationship between pain/disability and tissue injury, explaining the meaning of pain during exercises, and explaining the objectives of the implemented treatments.

SUMMARY:
The aim of this multicenter non-controlled study is to develop a multivariable prediction model of pain/disability improvements in patients with meniscal tears, after a physical therapy treatment based on therapeutic exercise and education.

DETAILED DESCRIPTION:
A multivariable prediction model for the improvement in shoulder pain and disability will be developed based on the following predictors:

* Body mass index [kg/m2, Fractional polynomials FP2].
* Smoking [Years, linear relationship].
* Employment status [3 categories].
* Maximum education degree [4 categories].
* Previous performance of physical exercise [2 categories].
* Baseline disability (measured with the Knee Injury and Ostoarthritis Outcome Score) [Fractional polynomials FP2].
* Baseline pain intensity (measured with a numeric pain rating scale) [Fractional polynomials FP2].
* Pain duration [Weeks, linear relationship]
* Pain catastrophizing (measured with the Pain Catastrophizing Scale) [Linear relationship].
* Patient's expectations (measured with the Musculoskeletal Outcomes Data Evaluation and Management System) [Linear relationship].

ELIGIBILITY:
Inclusion Criteria:

* Degenerative meniscal tears (medial and/or lateral), diagnosed by magnetic resonance imaging.
* Traumatic meniscal tears (medial and/or lateral), diagnosed by magnetic resonance imaging, originated 6 months ago or more.
* Pain intensity equal or greater to 3 points in a numeric pain rating scale, or a degree of disability in the KOOS questionnaire greater or equal to 15%.
* Pain lasting 3 months ore more.
* Adequate comprehension of written and spoken Spanish

Exclusion Criteria:

* Knee ligament injuries at the moment of recruitment.
* Presence of hip or ankle pathology that makes it impossible to peform knee therapeutic exercises.
* History of fracture in the lower limb within the last year.
* History of surgery in the lower lim within the last year.
* Presence of cancer, fibromyalgia, neurological and/or other systemic diseases.
* Cognitive impairment that makes it impossible to perform therapeutic exercise.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Knee disability | Baseline, change from baseline to 3-month, change from baseline to 6-month, and change from baseline to 1-year.
  Knee disability measured with the Knee Injury and Osteoarthritis Outcome Score, which ranges from 0 (no disability) to 100 (maximum degree of disability).

SECONDARY OUTCOMES:
Knee pain intensity | Baseline, change from baseline to 3-month, change from baseline to 6-month, and change from baseline to 1-year.
  Knee pain intensity measured with a numeric pain rating scale, which ranges from 0 (no pain) to 10 (worst imaginable pain).
Need for surgery | 3-month, 6-month, and 1-year.
  Need for surgery for the rotator cuff tear registered as a dichotomous variable (YES/NO).

OTHER OUTCOMES:
Pain Catastrophizing | Baseline
  Pain catastrophizing measured with the Pain Catastrophizing Scale, which ranges from 0 (minimum degree of catastrophizing) to 100 (maximum degree of catastrophizing).
Patient's expectations | Baseline
  Patient's expectations of improvement with therapeutic exercise measured with the Musculoskeletal Outcomes Data Evaluation and Management System, which ranges from 0 (minimum degree of expectations) to 100 (maximum degree of expectations).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
IPD data will be shared with other researchers upon reasonable request